CLINICAL TRIAL: NCT04556266
Title: A Phase I Trial Evaluating the Safety of Consolidative Infusions of CD19-Specific Chimeric Antigen Receptor (CAR) T Cells Following T-cell Depleted Allogeneic Transplantation for High Risk B-cell Malignancies
Brief Title: A Phase I Trial of Donor- Derived 19-28z CAR T Cells Following Allogeneic Transplant for the Treatment of CD19 Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No patients were enrolled to this study since being open to enrollment. Due to changes in available therapies, there aren't enough people who will be eligible for the study. Therefore, the study was closed.
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17-331
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2022-03

CONDITIONS: Leukemia; Lymphoma; Lymphoma, B-Cell
Keywords: Leukemia; Lymphoma; Lymphoma, B-Cell; Chimeric Antigen Receptor (CAR) T cells; CART cells; high-risk B-cell malignancies; 17-331; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Leukemia; Lymphoma; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort -1 (Experimental): Cohorts of 3-6 patients each will be treated with escalating doses of consolidative modified T cells at Day 30 (+/- 5 days) post allo-HSCT
  Total T-Cell Dose: 1 x 10^4 cells/kg
  Interventions: Biological: CAR T-Cell Infusion
- Cohort 1 (Experimental): Cohorts of 3-6 patients each will be treated with escalating doses of consolidative modified T cells at Day 30 (+/- 5 days) post allo-HSCT
  Total T-Cell Dose: 1 x 10^5 cells/kg
  Interventions: Biological: CAR T-Cell Infusion
- Cohort II (Experimental): Cohorts of 3-6 patients each will be treated with escalating doses of consolidative modified T cells at Day 30 (+/- 5 days) post allo-HSCT
  Total T-Cell Dose: 2 x 10^5 cells/kg
  Interventions: Biological: CAR T-Cell Infusion
- Cohort III (Experimental): Cohorts of 3-6 patients each will be treated with escalating doses of consolidative modified T cells at Day 30 (+/- 5 days) post allo-HSCT
  Total T-Cell Dose: 4 x 10^5 cells/kg
  Interventions: Biological: CAR T-Cell Infusion

INTERVENTIONS:
Biological: CAR T-Cell Infusion — Dose Level -1: 1 x 10^4 cells/kg Dose Level 1: 1 x 10^5 cells/kg Dose Level 2: 2 x 10^5 cells/kg Dose Level 3: 4 x 10^5 cells/kg

SUMMARY:
The purposed of this study is to determine whether an infusion with specialized 'modified T cells' (or CD19 chimeric antigen T cells, also called CD19 CAR T cells) that target the B cell marker will reduce the risk of relapse after transplant.

ELIGIBILITY:
Inclusion Criteria:

The following criteria must be met prior to the allogenic transplantation:

1. ALL in second remission or greater (≥ CR2)

   * Please refer to section 3.0 for more discussion of ALL in CR1 versus CR2
2. CLL

   1. High risk in any remission status as defined by 17p deletion or Richter's transformation, or
   2. All other patients eligible after at least 2 lines of standard or investigational chemotherapy
3. B-NHL

   1. Refractory or stable disease to last line of therapy per ICML 2014. Patients should have at least 2 lines of prior therapy.
   2. Relapsed disease in patients who are not candidates for autologous transplant
4. Patient's age is ≥ 18 and ≤ 60.
5. KPS ≥ 70%
6. Patients must have CD19 expression (by any detection method) demonstrated on their malignant cells at the time of enrollment on the protocol.
7. Patients relapsed after prior CD19 CAR T cell or blinatumomab are eligible for enrollment as long as CD19 expression is still prese on the malignant cells.
8. Patients who have a matched related donor willing to donate HSC for allograft and PBMC for CAR T cell generation
9. Patients must have adequate organ function measured by:

   1. Cardiac: asymptomatic or if symptomatic then LVEF at rest must be > 50%
   2. Hepatic: < 3x ULN ALT and < 1.5 total serum bilirubin, unless there is congenital benign hyperbilirubinemia.
   3. Renal: serum creatinine <1.3 mg/dl or if serum creatinine is outside the normal range, then CrCl > 60 ml/min (measured or calculated/estimated)
   4. Pulmonary: asymptomatic or if symptomatic, DLCO > 50% of predicted (corrected for hemoglobin)
   5. Negative serum pregnancy test for women of child-bearing potential is required

Exclusion Criteria:

1. Active and uncontrolled infection at time of transplantation. Please note that patients being actively treated for a viral reactivation may be enrolled on the protocol at the discretion of the investigators.
2. Patients who have undergone a prior allogeneic or autologous stem cell transplant within the previous six months.
3. Pregnant or breast feeding
4. HIV infection
5. Progressive disease at time of transplant
6. Patients with known autoimmune disease.
7. Patients with active or clinically significant neurological disorders, such as seizure disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 24 month
  To determine maximum tolerated dose (MTD) of intravenously administered allogeneic, donor-derived 19-28z CAR T cells administered following TCD allo-HSCT for patients with high-risk CD19+ malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Miguel-Angel Perales, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org